CLINICAL TRIAL: NCT01821482
Title: A Randomized Controlled Study of Dendritic and Cytokine-induced Killer Cells (DC-CIK) Treatment in Patients With Hepatocellular Carcinoma
Brief Title: A Study of DC-CIK to Treat Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Weiliang Sun, Investigator, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-01
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular carcinoma, DC-CIK
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): After complete resection or TACE, patients will receive 3 cycles of Dendritic and Cytokine-induced Killer Cells (DC-CIK) (every 4 weeks)
  Interventions: Biological: Dendritic and Cytokine-induced Killer Cells
- B (No Intervention): After complete resection or TACE, Patient only regularly follow up

INTERVENTIONS:
Biological: Dendritic and Cytokine-induced Killer Cells
  Other Names: DC-CIK
  Arms: A

SUMMARY:
The purpose of this study is to evaluate the efficacy of Dendritic and Cytokine-induced Killer Cells (DC-CIK) for hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
About 60 patients with HCC, who had received complete resection or TACE and got Complete remission (CR) or partial response (PR), will be randomly divided into group A (receive DC-CIK treatment) or group B (just regularly follow up), and the randomize ratio will be 1:1. Patients in group A will receive 2-3 cycles of DC-CIK cells treatment (every 4 weeks). Patients in group B will have no anti-tumor therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 18 years of age;
2. Hepatocellular carcinoma with histological or imaging and AFP diagnose, and had received complete resection or TACE and got CR or PR by imaging studies;
3. Patients who have a life expectancy of at least 12 weeks;
4. Eastern Cooperative Oncology Group (ECOG) performance status was 0 - 1;
5. The bone marrow functioned normally (WBC > 4.0×109/L, Hb > 120 g/L, PLT > 100×109/L);
6. The ECG results were normal, and the liver and kidney were functional.

Exclusion Criteria:

1. Patients who had distant metastases;
2. Patients with uncontrolled infection; underlying disease that was severe or life-threatening;
3. Patients who were pregnant or lactating;
4. ECOG perform status ≥ 2;
5. Patients who are suffering from auto immune diseases or patients who need to accept glucocorticoid treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(PFS) | 1 month

SECONDARY OUTCOMES:
Overall survival(OS) | 1 month
quality of life (QOL) | month

OTHER OUTCOMES:
Laboratory findings | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Hanfeng Liu, Study Chair — Guangxi Medical University
Locations (1):
- The first Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China